CLINICAL TRIAL: NCT03698188
Title: Evaluation of the Efficacy of Injectable Platelet-Rich Fibrin Versus Platelet-Rich Plasma in the Regeneration of Necrotic Immature Maxillary Anterior Teeth. (A Randomized Clinical Trial)
Brief Title: Comparative Evaluation of the Regenerative Capacity of Two Platelet Concentrates
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Maha Mohamed Abou-Heikal, assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 11888
Record Dates: First submitted 2018-10-03; First posted 2018-10-05 (Actual); Last update posted 2018-10-25 (Actual); Status verified 2018-10

CONDITIONS: Necrotic Pulp
MeSH Terms: conditions — Dental Pulp Necrosis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Injectable platelet-rich fibrin (Experimental): A platelet concentrate will be prepared from the patient's own blood in plain plastic tubes, without the use of anticoagulants, and applied immediately within the root canal before coagulation.
  Interventions: Procedure: Injectable platelet-rich fibrin
- Platelet-rich plasma (Active Comparator): A platelet concentrate will be prepared from the patient's own blood in tubes containing anticoagulants to maintain the fluid consistency and applied within the root canal.
  Interventions: Procedure: Platelet-rich plasma

INTERVENTIONS:
Procedure: Injectable platelet-rich fibrin — A blood sample will be drawn from the patient, centrifuged at 700 rpm for 3 minutes and the upper yellow fluid will be collected by a plastic syringe, avoiding the inclusion of the red blood cells underneath, and will be introduced within the root canal.
  Arms: Injectable platelet-rich fibrin
Procedure: Platelet-rich plasma — A blood sample will be drawn from the patient, centrifuged at 3000 rpm for 10 minutes and the upper yellow fluid will be collected by a plastic syringe, avoiding the inclusion of the red blood cells underneath, and will be introduced within the root canal.
  Arms: Platelet-rich plasma

SUMMARY:
Injectable platelet-rich fibrin (I-PRF) is a flowable blood concentrate that is entirely natural and allows ease of access and flow within the root canal. It was first developed in 2014 by modifying the centrifugation parameters. I-PRF has great potential in the field of endodontics. At present, it is still in its infancy and needs to be explored with regard to its regenerative efficacy.

To the best of our knowledge, this study is the first to clinically and comparatively investigate Platelet-rich plasma (PRP) and I-PRF.

DETAILED DESCRIPTION:
An ideal treatment option for an immature necrotic tooth is the regeneration of pulp-like tissue that is capable of boosting the continuation of normal root development. The use of platelet concentrates for that purpose is a clinically relevant, minimally invasive approach which has a promising potential of reducing the healing period. Among which, the most commonly employed is the Platelet-Rich Plasma that is not entirely natural. It involves the use of non-autologous anticoagulants such as bovine thrombin to maintain the fluid consistency which prevents clot formation and thus impairs wound healing, affects the coagulation process and can also trigger an immune reaction, thereby, suppressing regeneration.

PRP offers a short-term release of most of the growth factors unlike the Platelet-Rich Fibrin which allows for a more sustained release. PRF does not require any biochemical handling of blood and is easy to procure but due to the gel-like consistency, its adaptability within the root canal requires excessive removal of root dentin.

In addition, the application of recombinant growth factors within the root canal is associated with high cost which hinders its applicability in the common clinical practice.

Therefore, a new regenerative technique is required that combines the advantages of both PRP and PRF while overcoming their drawbacks.

ELIGIBILITY:
Inclusion Criteria:

* Patients having necrotic maxillary anterior tooth/teeth due to caries or trauma
* Radiographic criteria: preoperative radiograph showing incomplete root formation with a wide apical foramen.
* Positive patient/guardian compliance for participation in the study.

Exclusion Criteria:

* Uncooperative patient
* Lack of patient commitment to the treatment plan and the follow-up period
* Mature necrotic anterior teeth due to caries or trauma
* Vital maxillary anterior teeth with open apices
* Non-restorable teeth
* Grossly decayed or fractured teeth that require post and core as final restorations
* Presence of periodontal pockets
* Radiographically: presence of external or internal root resorption, fracture lines or cracks

Ages: 10 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 24 (Estimated)
Dates: Start 2018-11 (Estimated); Primary Completion 2019-05 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Increase in root length | one year follow-up
  root length will be measured on the preoperative and postoperative radiographs and the percentage increase in length will be calculated

SECONDARY OUTCOMES:
Restoration of tooth sensitivity | one year
  sensitivity will be measured by an electric pulp tester

CONTACTS AND LOCATIONS:
Overall Officials: Jealane El-Shafei, PhD, Study Director — Professor Doctor of Endodontics, Faculty of Dentistry, Cairo University.; Samia Shouman, PhD, Study Director — Professor Doctor of Medical Biochemistry, National Cancer Institute, Cairo University; Nehal Nabil, PhD, Study Director — Lecturer of Endodontics, Faculty of Dentistry, Cairo University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Varela HA, Souza JCM, Nascimento RM, Araujo RF Jr, Vasconcelos RC, Cavalcante RS, Guedes PM, Araujo AA. Injectable platelet rich fibrin: cell content, morphological, and protein characterization. Clin Oral Investig. 2019 Mar;23(3):1309-1318. doi: 10.1007/s00784-018-2555-2. Epub 2018 Jul 12. PMID 30003342
- [Background] Karde PA, Sethi KS, Mahale SA, Khedkar SU, Patil AG, Joshi CP. Comparative evaluation of platelet count and antimicrobial efficacy of injectable platelet-rich fibrin with other platelet concentrates: An in vitro study. J Indian Soc Periodontol. 2017 Mar-Apr;21(2):97-101. doi: 10.4103/jisp.jisp_201_17. PMID 29398852
- [Background] Wang X, Zhang Y, Choukroun J, Ghanaati S, Miron RJ. Effects of an injectable platelet-rich fibrin on osteoblast behavior and bone tissue formation in comparison to platelet-rich plasma. Platelets. 2018 Jan;29(1):48-55. doi: 10.1080/09537104.2017.1293807. Epub 2017 Mar 29. PMID 28351189
- [Background] Miron RJ, Fujioka-Kobayashi M, Hernandez M, Kandalam U, Zhang Y, Ghanaati S, Choukroun J. Injectable platelet rich fibrin (i-PRF): opportunities in regenerative dentistry? Clin Oral Investig. 2017 Nov;21(8):2619-2627. doi: 10.1007/s00784-017-2063-9. Epub 2017 Feb 2. PMID 28154995